CLINICAL TRIAL: NCT03703024
Title: A Double-blind, Randomized, Placebo-controlled Clinical Study to Evaluate the Efficacy of Raspberry Extract to Alleviate Symptoms of Osteoarthritis in the Knee
Brief Title: An Intervention Study Evaluating the Effects of a Raspberry Leaf Extract in an Osteoarthritic Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AFCRO-070
Record Dates: First submitted 2018-04-11; First posted 2018-10-11 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, placebo-controlled clinical study.
Who Masked: Participant, Investigator
Masking Description: Double blind model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo
- Low dose (Active Comparator): 200mg raspberry leaf extract. One capsule to be taken every morning over a 12-13 week period. Subjects will be instructed to take 1 capsule every morning with their breakfast.
  Interventions: Dietary Supplement: Raspberry Leaf Extract
- High dose (Active Comparator): 400mg raspberry leaf extract. One capsule to be taken every morning over a 12-13 week period. Subjects will be instructed to take 1 capsule every morning with their breakfast.
  Interventions: Dietary Supplement: Raspberry Leaf Extract

INTERVENTIONS:
Dietary Supplement: Raspberry Leaf Extract — Eligible subjects will be scheduled for an initial visit. The study will involve 3 visits over a 12 to 13-week period. One capsule to be taken every morning over a 12-13 week period.
  Arms: High dose; Low dose
Dietary Supplement: Placebo — Delivered in a capsule
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled clinical study to evaluate the efficacy of raspberry extract to alleviate symptoms of osteoarthritis in the knee.

DETAILED DESCRIPTION:
It is estimated that up to 260 subjects will be screened.

Subjects will undergo an initial phone screen and will be asked questions regarding their age, weight, and general health. Eligible subjects will be scheduled for an initial visit. The study will involve 3 visits over a 12 to 13-week period.

At the initial screening/baseline visit (Visit 1), the inclusion and exclusion criteria will be reviewed and the overall details of the study will be explained and informed consent obtained. Demographic data, vitals (blood pressure, heart rate and temperature), anthropometric measurements (weight, height and BMI) will be recorded. Family and medical history, and concomitant medications will be recorded. For women of child bearing age, a urine sample will be collected and pregnancy test performed. A blood sample (20mls) will be collected and haematology, biochemistry, glucose and hs-CRP will be measured. Additional serum will be aliquoted and stored and inflammatory biomarkers measured at a later date.

Subjects will complete the following questionnaires: International Physical Activity Questionnaire (IPAQ), Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale (WOMAC), Participant global assessment short form 36 (SF-36) and pain assessment using a Visual Analogue Scale (VAS).

Subjects will undergo the Short Physical Performance Battery (SPPB) test and will complete the 20-meter walk test.

Subjects will be provided with an electronic tablet and instructed to complete daily and record daily symptoms of pain (of the target knee), compliance in relation to taking the study product and record any rescue or other medication taken during the study duration.

Subjects will be randomised to one of three treatment groups as follows:

* Arm 1 -Placebo
* Arm 2 - 200mg raspberry extract
* Arm 3 - 400mg raspberry extract

Subjects will be provided with a box containing 6-weeks supply of study product, along with an additional 4-day supply in case of loss. Subjects will be instructed to take 1 capsule each morning, with their breakfast, for the duration of the study.

Subjects will return for visits at week 6 and week 12. At each visit the vitals, anthropometric measurements, concomitant medication and any adverse events will be recorded Subjects will complete the following questionnaires: International Physical Activity Questionnaire (IPAQ), Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale (WOMAC), Participant global assessment short form 36 (SF-36) and pain assessment using a Visual Analogue Scale (VAS).

Subjects will undergo the Short Physical Performance Battery (SPPB) test and will complete the 20-meter walk test.

Subjects will return their electronic device and the data will be downloaded and reviewed.

Subjects will return any unused study product and compliance will be assessed and new study product administered. On Visit 3, a blood sample (20mls) will be collected and haematology, biochemistry, glucose and hs-CRP will be measured. Additional serum will be aliquoted and stored and inflammatory biomarkers measured at a later date.

Subjects will be instructed to follow their standard diet and exercise routine and not consume medications that could interfere with the assessment of the study product for the duration of the study. Any symptoms and changes in their health status or medications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be aged 30 to 75 years (inclusive),
2. Be willing to provide informed consent,
3. Have a BMI between 18.5 and 32 kg/m2,
4. Have documented diagnosis of primary osteoarthritis (OA) of the target knee made at least 12 months prior to Screening,
5. Have radiographic evidence of OA in the tibio-femoral compartment of the target knee with at least 1 definite osteophyte and a measureable joint space, as diagnosed by standard X-rays taken no longer than 18 months,
6. Have mild to moderate pain not adequately or completely controlled with anti-inflammatory drugs,
7. Be able to perform the 20-meter walking test and to understand all questions from the WOMAC questionnaire.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Females are pregnant, lactating or wish to become pregnant during the study. Female subject is currently either of:

* non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation). (For purposes of this study, postmenopausal is defined as one year without menses), OR
* child bearing potential, the subject is eligible to enter and participate in this study if she is not lactating and has a negative urine pregnancy test at the screening visit, visit 2 and upon completion of the study at visit 5. The subject must also agree to one of the following methods of contraception: i. Complete abstinence from intercourse two weeks prior to administration of study drug, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where subject discontinues the study prematurely. (Subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit.) or, ii. Has a male sexual partner who is surgically sterilized prior to the Screen Visit and is the only male sexual partner for that subject or, iii. Sexual partner(s) is/are exclusively female or, iv. Oral contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. (Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 1 week following discontinuation of study medication).

  v. Use of double-barrier contraception, specifically, a spermicide plus a mechanical barrier (e.g. male condom, female diaphragm). The subject must be using this method for at least 1 week following the end of the study or, vi. Use of any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 2 weeks following the end of the study.
  1. Patient with secondary OA (due to a known disorder)
  2. Has modified Kellgren-Lawrence Numerical Grading System of grade IV in the patello-femoral compartment of the target knee confirmed by standard X-rays taken no longer than 12 months prior to Screening, and before any baseline assessment,
  3. Has clinically apparent tense effusion of the target knee or other joint,
  4. Has had viscosupplementation in any joint including the target knee or other joint within 9 months prior to Screening,
  5. Subject is taking any anti-inflammatory steroid medications, salicylates (aspirin) or Propionic acid derivatives (ibuprofen), for 2 weeks prior to study entry,
  6. Has concomitant inflammatory disease or other condition that affects the joints (e.g. rheumatoid arthritis, metabolic bone disease, psoriasis, gout, symptomatic chondrocalcinosis and active infection, etc.),
  7. Symptomatic OA of the contralateral knee that is not responsive to paracetamol and requires other therapy,
  8. Taking any calcium supplements (4-week washout) or other supplement e.g. glucosamine, chondroitin,
  9. Any medical condition deemed exclusionary by the Principal Investigator/Study doctor,
  10. Subject has a history of drug and / or alcohol abuse at the time of enrolment,
  11. Change of dietary habit within the preceding month,
  12. Subject with known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon and significant systemic disease,
  13. Subject currently involved in any other clinical trial or having participated in a trial within the preceding 90 days,
  14. Subject with known allergy to components of the test product,
  15. Subject has any concurrent medical or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements,
  16. Subject has a history of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years,
  17. Subject has a significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude supplement ingestion and/or assessment of safety and the study objectives,
  18. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation/severe, difficulty swallowing).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change, if any, in Pain Scores from baseline to the end of treatment using WOMAC | 12-13 weeks
  Change from baseline to study completion in pain scores on the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) To assess pain, stiffness, and physical function in patients with knee osteoarthritis
  The WOMAC consists of 24 items divided into 3 subscales:
  * Pain (5 items)
  * Stiffness (2 items)
  * Physical Function (17 items)
  The scale uses the following descriptors for all items: none, mild, moderate, severe, and extreme. These correspond to an ordinal scale of 0-4.
  The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Change, if any, from baseline to the end of treatment in WOMAC stiffness sub-score | 12-13 weeks
  WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) will be used to determine stiffness score.
  •Stiffness (2 items): after first waking and later in the day. The score for stiffness = 0-8. A higher score indicates stiffness.
Change, if any, from baseline to the end of treatment in WOMAC physical function sub-score. | 12-13 weeks
  WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) will be used to determine change in physical function from baseline to study completion.
  •Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties.
  The possible score for Physical function ranges from 0-68. A higher score indicates bad physical function.
Change, if any, from baseline to the end of treatment in WOMAC composite score | 12-13 weeks
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) will be used to determine a composite score of the 3 subscales.
Change, if any, in pain score using the VAS (for target knee joint & all other joints separately) | 12-13 weeks
  Visual Analogue Scale (VAS) features a horizontal line with the words NO PAIN on the left and WORST PAIN on the right. The subject marks the line to indicate overall pain in the previous 6 weeks. The line is then measured in mm and a higher measurement indicates greater pain.
Change in Quality of Life scores | 12-13 weeks
  Participant Global Assessment using a short form survey of 36 questions can observe subjects overall quality of life.
Change, if any, in walking speed | 12-13 weeks
  20 m walking test is timed at each visit and will be compared to determine if there is a change in speed throughout the duration of the study.
Change, if any, in physical performance | 12-13 weeks
  Short Physical Performance Battery (SPPB) is performed at each visit and will be compared to determine if there is a change in physical performance throughout the duration of the study. The SPPB includes a balance test, gait speed test and chair stand test. All of which can indicate if there is a change from week 1 to 12.
Change, if any, in activity levels | 12-13 weeks
  International Physical Activity Questionnaire (IPAQ) will be used to determine a change in activity levels throughout the duration of the study. Expressed as MET-min per week: MET level (walking, moderate/vigorous exercise) x minutes of activity/day x days per week.
Reduction in use of medication to manage pain compared to placebo | 12-13 weeks
  A device is provided to each subject upon randomisation with instructions to complete a series of questions daily. These questions include frequency and amount of medication consumed on said day. This is monitored to observe the use of medication throughout the 12-13 week study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Michael Molloy, Principal Investigator — Consultant Rheumatologist, Consultants Private Clinic, Cork University Hospital, Bishopstown road, Wilton, Cork.
Locations (1):
- Atlantia CRO, Heron House, Blackpool, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Henrotin Y, Cozannet RL, Fanca-Berthon P, Truillet R, Cohen-Solhal M, DunnGalvin G, Grouin JM, Doolan A. Rubus idaeus extract improves symptoms in knee osteoarthritis patients: results from a phase II double-blind randomized controlled trial. BMC Musculoskelet Disord. 2022 Jul 7;23(1):650. doi: 10.1186/s12891-022-05612-2. PMID 35799169
- See also: Kim LS, Axelrod LJ, Howard P, et al. Efficacy of methylsulfonylmethane (MSM) in osteoarthritis pain of the knee: a pilot clinical trial. Osteoarthritis and Cartilage. 2006 ; 14: 286-294. — https://www.ncbi.nlm.nih.gov/pubmed/16309928
- See also: Farid R, Mirfeizi Z, Mirheidari M, et al. Pycnogenol supplementation reduces pain and stiffness and improves physical function in adults with knee osteoarthritis. Nutrition Research. 2007; 27:692-697. — https://arizona.pure.elsevier.com/en/publications/pycnogenol-supplementation-reduces-pain-and-stiffness-and-improve
- See also: Belcaro G, Cesarone MR, Dugall M, et al. Product-evaluation registry of Meriva®, a curcumin phosphatidylcholine complex, for the complementary management of osteoarthritis. Panminerva Medica The Journal of the Italian Medical Association. 2010; 52:55-62. — http://accurateclinic.com/wp-content/uploads/2016/02/Product-evaluation-registry-of-Meriva%C2%AE-a-curcumin-phosphatidylcholine-complex-for-the-complementary-management-of-osteoarthritis-2010.pdf
- See also: Parsons M, Simpson M, Ponton T. Raspberry leaf and its effect on labour: safety and efficacy. Australian College of Midwives Incorporated Journal. 1999; 12:20-5. — https://www.ncbi.nlm.nih.gov/pubmed/10754818
- See also: Simpson M, Parsons M, Greenwood J, et al. Raspberry leaf in pregnancy: its safety and efficacy in labor. Journal of Midwifery & Women's Health. 2001; 46:51-9. — https://www.ncbi.nlm.nih.gov/pubmed/11370690
- See also: Nordeng H, Bayne K, Havnen GC, et al. Use of herbal drugs during pregnancy among 600 Norwegian women in relation to concurrent use of conventional drugs and pregnancy outcome. Complementary Therapies in Clinical Practice. 2011; 17:147-51. — https://www.ncbi.nlm.nih.gov/pubmed/21742280